CLINICAL TRIAL: NCT02092025
Title: Azilsartan Tablets Special Drug Use Surveillance: Long-term Use
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 279-011; JapicCTI-142441 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-02-26; First posted 2014-03-19 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azilsartan: Azilsartan 20 mg - 40 mg, tablet, orally, once daily for up to 12 months in participants based upon the disease severity. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Azilsartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan tablets
  Other Names: Azilva Tablets

SUMMARY:
The purpose of this survey is to evaluate the safety and efficacy of long-term use of azilsartan tablets (Azilva Tablets) in patients with hypertension in a routine clinical setting.

DETAILED DESCRIPTION:
This surveillance was designed to evaluate the safety and efficacy of long-term use of azilsartan tablets (Azilva Tablets) in hypertensive patients in daily medical practice.

The usual dosage for adult is 20 mg of azilsartan administered orally once daily. The dose can be adjusted according to the patient's age and condition. The maximum daily dose is 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients

Exclusion Criteria:

1. Patients with a history of hypersensitivity to any of the ingredients of Azilsartan
2. Patients who are pregnant or having possibilities of being pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 3437 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 738 investigative sites in Japan, from 20 June 2012 to 15 January 2016.
Pre-assignment Details: Participants with a historical diagnosis of hypertension were enrolled to receive Azilsartan 20 milligram (mg) - 40 mg tablet, orally, once daily for up to 12 months.
Period: Overall Study
Arm/Group | Azilsartan
Started | 3437
Completed | 3369
Not Completed | 68
Not completed — Case Report Forms Uncollected | 44
Not completed — Protocol Deviation | 24

BASELINE CHARACTERISTICS:
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Azilsartan
Number analyzed (Participants) | 3369
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1690
  Male | 1679
Region of Enrollment [Number; unit: Participants]
  Japan | 3369
Weight [Mean (Standard Deviation); unit: kg] — Population: The number analyzed is the number of participants with data available for analysis.
  kg
    number analyzed (Participants) | 2396
    (all) | 60.81 (13.716)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]. Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 2261
    (all) | 24.27 (4.096)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 3291
    Inpatient | 78
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had no Presence of Medical Complications | 956
    Had Presence of Medical Complications | 2413
Estimated Glomerular Filtration Rate (eGFR) [Count of Participants; unit: Participants]
  < 15 mL/min/1.73 m^2 | 61
  ≥ 15 mL/min/1.73 m^2 and < 30 mL/min/1.73 m^2 | 45
  ≥ 30 mL/min/1.73 m^2 and < 45 mL/min/1.73 m^2 | 184
  ≥ 45 mL/min/1.73 m^2 and < 60 mL/min/1.73 m^2 | 390
  ≥ 60 mL/min/1.73 m^2 and < 90 mL/min/1.73 m^2 | 1198
  ≥ 90 mL/min/1.73 m^2 | 288
  Unknown | 1203
Drinking Habits [Count of Participants; unit: Participants]
  Current Drinker | 828 (20.43)
  Not Current Drinker | 1823
  Unknown | 718
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 1572 (14.25)
  Current Smoker | 396
  Ex-Smoker | 539
  Unknown | 862
Clinical Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — Population: The number analyzed is the number of participants with data available for analysis.
  mmHg
    number analyzed (Participants) | 3359
    (all) | 155.1 (20.43)
Clinical Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 3359
    (all) | 86.7 (14.25)
SBP/DBP Classification [Count of Participants; unit: Participants]
  SBP < 140 mmHg and DBP < 90 mmHg | 552
  SBP ≥ 140 mmHg and DBP ≥ 90 mmHg | 2807
  Not Measured | 10
Pulse Rate [Mean (Standard Deviation); unit: bpm] — Population: The number analyzed is the number of participants with data available for analysis.
  bpm
    number analyzed (Participants) | 2983
    (all) | 74.1 (10.99)
Taking Hypertension Drug in 2 Months Before Baseline [Count of Participants; unit: Participants]
  Had Not Taken | 1080
  Had Taken | 2289

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to 12 Months
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan
Number analyzed (Participants) | 3369
Participants | 94

2. Secondary Outcome: Changes From Baseline in Systolic Blood Pressure (SBP) at Each Time Point
Description: Reported data are changes in SBP from baseline at Month 1 and final assessment (up to 12 months).
Time Frame: Baseline, Month 1 and final assessment (up to 12 Months)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'n' is number of participants analyzed at the given time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 3359
mmHg
  Change in SBP at Month 1: number analyzed (Participants) | 2895
  Change in SBP at Month 1 | -15.4 (19.99)
  Change in SBP at Final Assessment: number analyzed (Participants) | 3240
  Change in SBP at Final Assessment | -19.8 (22.80)

3. Secondary Outcome: Changes From Baseline in Diastolic Blood Pressure (DBP) at Each Time Point
Description: Reported data are changes in DBP from baseline at Month 1 and final assessment (up to 12 months).
Time Frame: Baseline, Month 1 and Final assessment (up to 12 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 3359
mmHg
  Change in DBP at Month 1: number analyzed (Participants) | 2895
  Change in DBP at Month 1 | -7.7 (12.55)
  Change in DBP at Final Assessment: number analyzed (Participants) | 3240
  Change in DBP at Final Assessment | -10.3 (13.91)

ADVERSE EVENTS:
Time Frame: Up to 12 Month
Description: Investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only non-serious ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Azilsartan
Serious Adverse Events (participants affected / at risk) | 10/3369
Other Adverse Events (participants affected / at risk) | 15/3369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan (N=3369)
Decreased appetite (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Asthenia (General disorders) | 1
Drowning (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan (N=3369)
Dizziness (Nervous system disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.